CLINICAL TRIAL: NCT00787774
Title: Integrase Resistance Analysis in Treated Experienced HIV Patients Who Interrupted Raltegravir Due to Incomplete Viral Suppression
Brief Title: Integrase Resistance Analysis in HIV Patients Who Interrupted Raltegravir Due to Incomplete Viral Suppression
Acronym: RAL-dyn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: José Luis Blanco Arévalo, Hospital Clínic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RAL-dyn
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: HIV Infection
Keywords: HIV; resistance; integrase
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: resume raltegravir — resume raltegravir after 16 weeks of stopping

SUMMARY:
Prospective study to evaluate the potential persistent viral effect of raltegravir in 20 treatment experienced HIV patients with incomplete viral suppression

ELIGIBILITY:
Inclusion Criteria:

* Subjects on Raltegravir-containing regimen with confirmed virological failure (VL >500c/mL for > 3 months).
* Patients treated with a raltegravir-containing regimen for at least for 24 weeks.
* CD4 cell count > 50 cell/mm3.
* Adherence >90%, measured by short -self report questionnaire during the 3 months preceding the study entry.
* No reasonable additional therapeutic options

Exclusion Criteria:

* History or suspicion of alcohol or drug use which in the investigator's opinion would likely compromise subjects' safety and/or study procedures.
* A positive urine drug test for amphetamines, cocaine and opioids at two consecutive screenings (a positive drug test at study screening will be repeated at baseline).
* Life expectancy less than 6 months.
* Subject has any currently active AIDS defining illness (Category C conditions according to the CDC Classification System for HIV Infection 1993) with the following 2 exceptions:

  1. Stable cutaneous Kaposi's Sarcoma that is unlikely to require any form of systemic therapy during the study period.
  2. Wasting syndrome due to HIV infection if, in the investigator's opinion, it is not actively progressive.
* Any active clinically significant disease (e.g. TB, cardiac dysfunction) or findings during screening of medical history or physical examination that in the investigator's opinion, would compromise the outcome of the study.
* Pregnant or breast-feeding female.
* Renal impairment: serum creatinine > 2 x ULN.
* Chronic Hepatitis B or C with ALT or AST > 3 x ULN.
* Acute Hepatitis A, B or C. Acute Hepatitis A, B or C.
* Any grade 3 or 4 toxicity according to the enhanced ACTG grading severity list, except for grade 3 or 4 asymptomatic triglyceride/cholesterol elevations, isolated grade 3 increased in GGT, grade 3 increases in glucose, asymptomatic grade 3 increases in amylase with no elevation of lipase.
* Currently significant diarrhea, gastric stasis or constipation that in the investigator's opinion could influence drug absorption or bioavailability.
* Subjects with clinical or laboratory evidence of significantly decreased hepatic function or decompensation, irrespective of liver enzyme levels (INR > 1.3 or albumin < 30g/l or bilirubin > 2.5 x ULN).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Change in viral load after resuming raltegravir in patients with incomplete viral suppression with raltegravir. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Gatell, MD, Study Chair — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Barcelona, Spain